CLINICAL TRIAL: NCT07095088
Title: Effects of Awareness-based Parenting and Birth Preparation Education Given to Couples on Materna-paternal Bonding, Birthparameters and Postpartum Harmony
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MERVE GÜL TİREN, Responsible Party Type: Principal Investigator, PhD student Name: Merve Gül Tiren, Kayseri Training and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kayseri city hospital
Record Dates: First submitted 2025-06-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mindfulness; Mindfulness Based Stress Reduction
Keywords: birth; childbirth preparation classes; mindfulness; mbcp
MeSH Terms: interventions — Mind-Body Therapies

STUDY DESIGN:
Intervention Model Description: In this study, the experimental design of the quantitative research method was used. Quantitative research is a research that includes the process of observing and measuring numerical values objectively and systematically in order to obtain information about the current situation and facts, and the measurements can be repeated. Quantitative research focuses on the relationships and differences between variables, makes predictions about the future and has the aim of generalization. In quantitative research based on the positivism approach, hypotheses are clearly determined and tested. Since the research examined the effects of the awareness-based parenting and birth preparation training given in the birth preparation class on maternal-paternal attachment, birth parameters and postpartum sleep of a sample group that reached the power to represent the universe, the experimental design with a pre-test and post-test control.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Childbirth and Parenting (MBCP) (Experimental): 9 weeks of MBCP training will be provided.In addition to the 1-week birth preparation training at the Pregnancy School of Kayseri City Education and Research Hospital, the intervention group received Mindfulness-Based Parenting and Birth Preparation Training. This training aimed to teach participants how to monitor their thoughts and emotional states, how to deepen their sensory awareness of their bodies, how to be more careful about how their minds work, and how to deepen their sensory self-awareness, so that they would be more sensitive during the birth and parenting processes. A total of 9 separate sessions were implemented. Mindfulness-Based Parenting and Birth Preparation Training was held once a week for 9 weeks, with the duration of each session varying according to the parents' compliance and needs in the program, and each session lasted an average of 150 minutes.
  Interventions: Other: Mind-body therapy
- clasical education (No Intervention): No additional training was given to the control group other than the 1-week birth preparation training at the Kayseri City Training and Research Hospital Pregnancy School.

INTERVENTIONS:
Other: Mind-body therapy — In addition to the 1-week birth preparation training at the Kayseri City Education and Research Hospital Pregnancy School, the intervention group received Mindfulness-Based Parenting and Birth Preparation Training. This training aimed to teach participants how to monitor their thoughts and emotional states, how to deepen their sensory awareness of their bodies, how to be more careful about how their minds work, and how to deepen their sensory self-awareness, so that they would be more sensitive during the birth and parenting processes. A total of 9 separate sessions were implemented. Mindfulness-Based Parenting and Birth Preparation Training was held once a week for 9 weeks, with the duration of each session varying according to the parents' compliance and needs in the program, and each session lasted an average of 150 minutes.
  Arms: Mindfulness-Based Childbirth and Parenting (MBCP)

SUMMARY:
Nurses, who play a key role in maternal and infant health, take action with evidence-based practices to reduce fear of childbirth, encourage natural birth, and improve negative pre-pregnancy, pregnancy, and post-pregnancy outcomes caused by fear.Considering the increasing rates of elective cesarean sections in developed countries, interventions against fear of childbirth have become more important. The negative effects of cesarean section on both maternal and infant health and the damage it causes to the health system due to increased costs are clear . For all these reasons, the inclusion of awareness-based interventions such as MBCP in childbirth preparation class education programs not only aims to reduce the increasing cesarean section rates, but also aims to provide awareness that women and their partners can benefit from not only during pregnancy, birth, and parenthood, but throughout their lives.

DETAILED DESCRIPTION:
According to the Turkish Language Association, the word parent means mother and father. It is also described as a nuclear family and represents the mother and father of a child . The meaning of being a parent is defined as the continuous provision of care, needs and support for a child for development and survival .

Becoming a parent is one of the developmental transition periods that include radical changes and add new roles and responsibilities to an individual's life . This process of change is called the transition to parenthood. Although there are many different views on when the transition to parenthood begins and ends, the most widely accepted view is that it begins with pregnancy for individuals who become mothers/fathers for the first time and ends within a few months after birth. The transition period is followed by the parenthood period .

The transition period to parenthood also brings about parent-infant bonding. The term attachment refers to the ability to establish and maintain an emotionally positive, mutual, and supportive relationship between babies and parents. If the relationship is established appropriately, adults adapt themselves to their babies and babies give adults clues about their needs. This relationship, which develops in the early period, has an important place in the physical, psychological, and intellectual development of the child and continues to be effective throughout life. The family-baby bonding process develops in three periods: pregnancy, birth, and postpartum . During pregnancy, it is important for parents to feel and caress their baby physically, to believe that their baby is in touch with them, to talk to the fetus, to say its name, to think about their baby, to feel positive feelings about their baby, and to imagine their baby's future situation in terms of the development of attachment . It is stated that the attachment that begins during pregnancy gradually increases as the pregnancy progresses and strengthens after the baby is born .In a study examining attachment, it was determined that there was a strong and significant relationship between prenatal attachment and postpartum attachment . Since the conscious emotions created by attachment are motivating during pregnancy and facilitate adaptation to the parenting role, they also positively affect the parent-infant adaptation process . The pregnancy period is seen as an important preparation period in which physiological, psychological, social and emotional changes are experienced for parenthood and adaptation to these changes is required. Especially individuals who will become mothers and fathers for the first time may experience some feelings of uncertainty regarding the changes experienced during pregnancy, birth and the postpartum period. Parents want the pregnancy process to be smooth, the birth to be painless and with high satisfaction . However, during this process, they experience complex emotions such as anxiety, fear, and excitement. Fears usually arise from the possibility of an episiotomy during vaginal birth, the possibility of a tear in the perineum, the pain felt during all these processes, and the responsibilities of being a parent regarding baby care . There are many educational programs that focus on attitudes and behaviors for parents in order to facilitate individuals' adaptation to these changes and to better manage their transition to parenthood. These programs have a positive effect on the individual well-being of parents, their ability to acquire parenting skills in a healthy way, and the healthy development of the child . By supporting the uncertainty of this transition process with educational programs in the prenatal period, family-baby bonding and adaptation can be achieved, and pregnancy, birth and postpartum processes can be continued in a healthy way One of the behavioral intervention programs used to adapt to the changes experienced during pregnancy, birth and postpartum and to continue the transition to parenthood in a healthy way is Conscious Awareness-Based Applications. Conscious awareness is an experiential process in which attention is directed purposefully and consciously to what is happening in the body and mind at that moment, and the content that emerges as a result of these observations is accepted with curiosity, understanding and compassion without judgment, analysis or reaction. According to the Turkish Language Association, the word parent means mother and father. It is also described as a nuclear family and represents the mother and father of a child . The meaning of being a parent is defined as the continuous provision of care, needs and support for a child for development and survival .

Becoming a parent is one of the developmental transition periods that include radical changes and add new roles and responsibilities to an individual's life This process of change is called the transition to parenthood . Although there are many different views on when the transition to parenthood begins and ends, the most widely accepted view is that it begins with pregnancy for individuals who become mothers/fathers for the first time and ends within a few months after birth. The transition period is followed by the parenthood period .

The transition period to parenthood also brings about parent-infant bonding. The term attachment refers to the ability to establish and maintain an emotionally positive, mutual, and supportive relationship between babies and parents. If the relationship is established appropriately, adults adapt themselves to their babies and babies give adults clues about their needs. This relationship, which develops in the early period, has an important place in the physical, psychological, and intellectual development of the child and continues to be effective throughout life. The family-baby bonding process develops in three periods: pregnancy, birth, and postpartum. During pregnancy, it is important for parents to feel and caress their baby physically, to believe that their baby is in touch with them, to talk to the fetus, to say its name, to think about their baby, to feel positive feelings about their baby, and to imagine their baby's future situation in terms of the development of attachment .It is stated that the attachment that begins during pregnancy gradually increases as the pregnancy progresses and strengthens after the baby is born . In a study examining attachment, it was determined that there was a strong and significant relationship between prenatal attachment and postpartum attachment . Since the conscious emotions created by attachment are motivating during pregnancy and facilitate adaptation to the parenting role, they also positively affect the parent-infant adaptation process. The pregnancy period is seen as an important preparation period in which physiological, psychological, social and emotional changes are experienced for parenthood and adaptation to these changes is required. Especially individuals who will become mothers and fathers for the first time may experience some feelings of uncertainty regarding the changes experienced during pregnancy, birth and the postpartum period. Parents want the pregnancy process to be smooth, the birth to be painless and with high satisfaction .However, during this process, they experience complex emotions such as anxiety, fear, and excitement . Fears usually arise from the possibility of an episiotomy during vaginal birth, the possibility of a tear in the perineum, the pain felt during all these processes, and the responsibilities of being a parent regarding baby care .There are many educational programs that focus on attitudes and behaviors for parents in order to facilitate individuals' adaptation to these changes and to better manage their transition to parenthood. These programs have a positive effect on the individual well-being of parents, their ability to acquire parenting skills in a healthy way, and the healthy development of the child. By supporting the uncertainty of this transition process with educational programs in the prenatal period, family-baby bonding and adaptation can be achieved and pregnancy, birth and postpartum processes can be continued in a healthy way . It is a skill that allows us not to be passive towards everything that is happening in the moment and is associated with reducing all levels of suffering and increasing our well-being with all our positive, negative and neutral experiences. Due to the stated effects, these interventions are important for parents to develop awareness and acceptance of thoughts, feelings and body sensations, reduce reactivity, avoid disturbing experiences, accept the roles and responsibilities of parenting in a non-judgmental manner, learn to use mechanisms to cope with the stress of parenting and show compassion to themselves and their children.

Mindfulness-based training can be integrated into childbirth preparation training as it is a method that can be used to improve birth parameters. When the literature is examined, there are studies examining the effects of Mindfulness-Based Parenting and Childbirth Preparation Training (MBCP) on mothers in the perinatal period, but there are limited studies that include fathers in the practice and studies examining the relationship between mindfulness training and adaptation and attachment. It is stated that actively including both parents in group-based parenting training is more effective in increasing the efficiency of the program . Meleis stated that mindfulness is an important feature of the transition. The higher the awareness of the individual regarding the new role that he/she will undertake at the end of the transition, the higher the level of competence and success in the role will be . Therefore, MBCP training implemented during the transition to parenthood is important as it will increase competence and adaptation to parenting roles, facilitate the birth process, and ensure maternal and paternal bonding, and increase the quality of pregnancy, birth, and postpartum care. In this context, it is thought that this study will serve the article stated in the 12th Development Plan (2024-2028) that "Starting from the prenatal period, services regarding children's health, nutrition, early learning, responsive and sensitive care, safe environment, and social protection policies will be provided, and their accessibility will be increased and their quality will be improved" . In this context, it is expected that MBCP training will affect the behavioral changes of parents. Parents will be able to easily access the trainings and will be able to integrate the awareness-based practices they learn in the training into every moment of their lives and parenting roles and make them sustainable.

For all these reasons, this research was planned to investigate the effects of the Awareness-Based Parenting and Birth Preparation Training given to couples on maternal-paternal bonding, birth parameters and postpartum sleep. It is thought that the trainings that parents receive with awareness of their own bodies and the birth process will positively contribute to the pregnancy, birth and postpartum process. In this way, it is aimed that this training activity organized for the purpose of having a healthy birth will contribute to the third goal of Sustainable Development, "Securing Healthy and Quality Life at All Ages" and that the expectant mothers will have a healthier birth and develop awareness about acting considering the health of the mother and baby during pregnancy, birth and postpartum processes .

The research question was formed as "What is the effect of the Awareness-Based Parenting and Birth Preparation Training on maternal-paternal bonding, birth parameters and postpartum sleep?"

ELIGIBILITY:
Inclusion criteria:

* Women aged 18-35,
* Women in their first pregnancy,
* Women in their 24-28th weeks of pregnancy,
* Women accepted to Pregnancy School training during the study period,
* Women with at least a literate education level, and
* Women without a communication barrier were included in the study.

Exclusion Criteria:

- • Women with psychiatric disorders,

* Women with pregnancy-related risk factors that could lead to a risk of preterm birth,
* Women with chronic illnesses that could lead to a risk of preterm birth were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women and their spouses participated in the application
Enrollment: 24 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Mindful Attention Awareness Scale(MAAS) total score to assess change in trait mindfulness | Baseline (pre-intervention) and post-intervention (week 8)
  The MAAS is a 15-item self-report questionnaire developed by Brown & Ryan (2003) and adapted into Turkish by Özyeşil et al. (2011). It measures the frequency of mindful states in daily life using a 6-point Likert scale (1 = Almost always to 6 = Almost never), with total scores ranging between 15 and 90. Higher scores reflect higher dispositional mindfulness.
  Unit of Measure:
  Total Score (15-90)

SECONDARY OUTCOMES:
Wijma Delivery Expectancy Questionnaire (W-DEQ)total score to assess fear of childbirth | Baseline (gestational week 28-30) and post-intervention (gestational week 36)
  The W-DEQ is a 33-item self-report questionnaire developed by Wijma et al. (1998) to assess fear of childbirth. Items are scored on a 6-point Likert scale (0 = Not at all to 5 = Extremely), with total scores ranging from 0 to 165. Higher scores indicate greater fear. The Turkish version has been validated in pregnant populations.
  Unit of Measure:
  Total Score (range: 0-165)
Visual Analog Scale (VAS)score to assess perceived labor pain | IMMEDIATELY AFTER BIRTH
  Pain intensity will be measured using the Visual Analog Scale (VAS), a self-reported measure where participants rate their pain on a scale from 0 (no pain) to 10 (worst imaginable pain). The score reflects the subjective intensity of labor pain during active labor. VAS is a widely used and validated tool for assessing acute pain.
  Unit of Measure:
  Score (range: 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Şehir Hastanesi, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
güvenlikle ilgili şüphelerim var

REFERENCES:
- See also: Related Info — https://www.mindfulnessinstitute.com.tr/mindfulness-nedir

DOCUMENTS (1):
  • Study Protocol (2025-06-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT07095088/Prot_000.pdf